CLINICAL TRIAL: NCT02288559
Title: A Phase II, Multicenter, Randomized, Single-Masked, Sham Injection-Controlled Exposure-Response Study of Lampalizumab Intravitreal Injections Administered Every Two Weeks or Every Four Weeks to Patients With Geographic Atrophy
Brief Title: A Study of Lampalizumab Intravitreal Injections Administered Every Two Weeks or Every Four Weeks to Participants With Geographic Atrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GX29455
Record Dates: First submitted 2014-11-07; First posted 2014-11-11 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy | interventions — salicylhydroxamic acid; lampalizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Lampalizumab: Open-label Safety Run-In (Experimental): Participants will receive 10 milligrams (mg) lampalizumab intravitreally Q2W during the safety run-in period.
  Interventions: Drug: Lampalizumab
- Q2W Lampalizumab: Randomized Treatment (Experimental): Participants will receive 10 mg dose of lampalizumab intravitreally Q2W during the 24-week treatment period.
  Interventions: Drug: Lampalizumab
- Q4W Lampalizumab: Randomized Treatment (Experimental): Participants will receive 10 mg dose of lampalizumab intravitreally Q4W during the 24-week treatment period.
  Interventions: Drug: Lampalizumab
- Sham: Randomized Treatment (Sham Comparator): Participants randomized to control arms will receive sham injections, that mimics intravitreal injection of lampalizumab.
  Interventions: Other: Sham

INTERVENTIONS:
Other: Sham — Sham injection will be administered as a matching intravitreal injection of lampalizumab.
  Arms: Sham: Randomized Treatment
Drug: Lampalizumab — 10 mg dose of lampalizumab administered intravitreally
  Arms: Lampalizumab: Open-label Safety Run-In; Q2W Lampalizumab: Randomized Treatment; Q4W Lampalizumab: Randomized Treatment

SUMMARY:
This multicenter, randomized, single-masked, sham injection-controlled study will investigate the exposure-response and safety of lampalizumab administered intravitreally every 2 weeks (Q2W) or every 4 weeks (Q4W) for 24 weeks in participants with geographic atrophy (GA) secondary to age-related macular degeneration (AMD). A safety run-in assessment will be conducted prior to initiating enrollment in the randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Complement Factor I (CFI) profile biomarker-positive result
* Women of child bearing potential and men should remain abstinent or use contraceptive methods

Exclusion Criteria:

* History of vitrectomy surgery, submacular surgery, or other surgical intervention for AMD in study eye
* Previous subfoveal focal laser photocoagulation in study eye
* Laser photocoagulation in the study eye
* Prior treatment with external-beam radiation therapy or transpupillary thermotherapy in study eye
* Previous intravitreal drug administration in study eye. A single intraoperative administration of a corticosteroid during cataract surgery at least 3 months prior to screening is permitted
* Previous cell-based intraocular treatment in study eye
* Intraocular surgery in study eye
* Uncontrolled glaucoma and history of glaucoma-filtering surgery in study eye
* History of corneal transplant in study eye
* GA in either eye due to causes other than AMD
* Proliferative diabetic retinopathy in either eye
* Active or history of neovascular (wet) AMD in either eye
* History of idiopathic or autoimmune-associated uveitis, ocular or intraocular conditions, and infectious or inflammatory ocular disease
* Active uveitis and infectious conjunctivitis, keratitis, scleritis or endophthalmitis
* Previous systemic treatment with complement inhibitor and with inhibitors/modulators of visual cycle
* Previous expression vector mediated intraocular treatments
* Uncontrolled blood pressure and atrial fibrillation
* Medical conditions associated with clinically significant risk for bleeding-
* Predisposition or history of increased risk for infection
* Active malignancy within the previous 12 months except for appropriately treated carcinoma in situ of cervix, resolved non-melanoma skin carcinoma, and prostate cancer with a Gleason score of less than or equal to 6, and a stable prostate-specific antigen for greater than or equal to (>/=) 12 months
* History of severe allergic reaction or anaphylactic reaction to a biologic agent or known hypersensitivity to any component of lampalizumab injection
* Women of child bearing potential must have a negative serum pregnancy test within 28 days prior to initiation of study treatment
* Previous participation in other studies of investigational drugs

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (36):
- United States (36):
  - Barnet Dulaney Perkins Eye Center, Mesa, Arizona
  - University of Arizona; Banner University Medical, Department of Opthalmology, Tucson, Arizona
  - Northwest Arkansas Retina Associates, Springdale, Arkansas
  - Retinal Diagnostic Center, Campbell, California
  - The Retina Partners, Encino, California
  - Loma Linda University, Loma Linda, California
  - San Diego Retina Associates, Oceanside, California
  - West Coast Retina Medical Group, San Francisco, California
  - California Retina Consultants, Santa Barbara, California
  - Colorado Retina Associates, PC, Golden, Colorado
  - Florida Eye Microsurgical Inst, Boynton Beach, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Retina Care Specialists, Palm Beach Gardens, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Elman Retina Group, Baltimore, Maryland
  - Vitreoretinal Surgery, Edina, Minnesota
  - The Retina Institute, St Louis, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - Eye Associates of New Mexico, Albuquerque, New Mexico
  - Western Carolina Retinal Associate PA, Asheville, North Carolina
  - Char Eye Ear &Throat Assoc, Charlotte, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Retina Assoc of Cleveland Inc, Cleveland, Ohio
  - Dean McGee Eye Institute, Oklahoma City, Oklahoma
  - Retina Cons of Charleston, Charleston, South Carolina
  - Carolina Retina Center PA, Columbia, South Carolina
  - Charles Retina Institution, Germantown, Tennessee
  - Southeastern Retina Associates, Knoxville, Tennessee
  - Tennessee Retina PC., Nashville, Tennessee
  - W Texas Retina Consultants PA, Abilene, Texas
  - Texas Retina Associates, Dallas, Texas
  - Retina Specialists, DeSoto, Texas
  - Wagner Macula & Retina Center, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 332 participants were screened and 92 participants were randomized out of which 3 participants from one site were removed from the randomized population due to serious good clinical practice (GCP) noncompliance. Out of 89, 4 participants were excluded from the randomized population as they did not have any post-baseline measurement.
  .
Groups:
- Sham Q2W: Participants received sham comparator Q2W (once every 2 weeks) for 24 weeks.
- Sham Q4W: Participants received sham comparator Q4W (once every 4 weeks) for 24 weeks.
- Lampalizumab Q2W: Participants received 10 milligrams (mg) dose of lampalizumab administered by intravitreal injections Q2W for 24 weeks.
- Lampalizumab Q4W: Participants received 10 mg dose of lampalizumab administered by intravitreal injections Q4W for 24 weeks.
Period: Overall Study
Arm/Group | Sham Q2W | Sham Q4W | Lampalizumab Q2W | Lampalizumab Q4W
Started | 10 | 11 | 46 | 22
Completed | 9 | 10 | 35 | 20
Not Completed | 1 | 1 | 11 | 2
Not completed — Adverse Event | 1 | 1 | 5 | 0
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1
Not completed — Reason Not Specified | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) population included participants who were randomly assigned to study treatment and had at least one post-baseline geographic atrophy (GA) area measurement.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Q2W | Sham Q4W | Lampalizumab Q2W | Lampalizumab Q4W | Total
Number analyzed (Participants) | 10 | 10 | 43 | 22 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.4 (4.4) | 78.2 (7.7) | 78.3 (8.0) | 80.1 (7.7) | 78.2 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 25 | 9 | 49
  Male | 3 | 2 | 18 | 13 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 10 | 10 | 42 | 22 | 84
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 1 | 0 | 2
  White | 9 | 9 | 42 | 22 | 82
Geographic Atrophy Area, as Assessed by Fundus Autofluorescence (FAF) [Mean (Standard Deviation); unit: millimeter square (mm^2)] — GA or the death of photoreceptors and surrounding cells in the retina, is a common condition in participants with age-related macular degeneration (AMD). The death of these photoreceptors results in lesions that cause vision loss. The change in GA lesion area was measured by FAF and analysis of FAF images was performed by the central reading center.
  millimeter square (mm^2) | 7.034 (2.747) | 6.891 (3.050) | 8.755 (4.059) | 7.172 (4.192) | 7.923 (3.894)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Geographic Atrophy (GA) Area, as Assessed by Fundus Autofluorescence (FAF) at Week 24
Description: GA or the death of photoreceptors and surrounding cells in the retina, is a common condition in participants with age-related macular degeneration (AMD). The death of these photoreceptors results in lesions that cause vision loss. The change in GA lesion area was measured by FAF and analysis of FAF images was performed by the central reading center. A positive change from baseline indicates an increase in size of geographic atrophy lesion area (worsening; disease progression). BCVA=best corrected visual acuity; ETDRS=Early Treatment Diabetic Retinopathy Scale.
Time Frame: Baseline, Week 24
Population: Modified intent-to-treat (mITT) population included participants who were randomly assigned to study treatment and had at least one post-baseline GA area measurement. Number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Mean (Standard Error); unit: mm^2
Arm/Group | Sham Q2W | Sham Q4W | Lampalizumab Q2W | Lampalizumab Q4W
Number analyzed (Participants) | 10 | 10 | 43 | 22
mm^2 | 0.614 (0.188) | 1.121 (0.179) | 1.049 (0.094) | 0.911 (0.123)
Statistical Analysis 1: Comparison: Sham Q2W vs Lampalizumab Q2W; Test type: Superiority; p = 0.0428, Mixed-Effect Model Repeated Measures; MMRM analysis variables: treatment group, visit, treatment-by-visit interaction, baseline GA area, and BCVA ETDRS chart Snellen equivalent category; Difference in Adjusted Means = 0.435, 80% CI 2-sided [0.162 to 0.707]
Statistical Analysis 2: Comparison: Sham Q4W vs Lampalizumab Q4W; Test type: Superiority; p = 0.3361, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in Adjusted Means = -0.210, 80% CI 2-sided [-0.491 to 0.071]

2. Secondary Outcome: Serum Concentrations of Lampalizumab (Q2W)
Description: Lower than reportable (LTR) results on pre-dose sample were set to 0, and LTR results on post-dose sample were set to half of lower limit of quantification (LLOQ) (0.5 nanograms per milliliter (ng/mL)).
Time Frame: Baseline (Day 1, predose and postdose), Weeks 2,4,8,16 and 24, early termination, unscheduled predose and postdose
Population: Pharmacokinetics (PK) population included participants randomized to lampalizumab treatment who received at least one dose of study drug and provided at least one serum sample for determination of lampalizumab. Number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Lampalizumab Q2W
Number analyzed (Participants) | 46
ng/mL
  Day 1 (Predose): number analyzed (Participants) | 43
  Day 1 (Predose) | NA (NA) — Geometric mean and geometric coefficient of variation were not calculable as more than one-third of the values were LTR.
  Day 1 (Postdose): number analyzed (Participants) | 44
  Day 1 (Postdose) | 1.31 (NA) — Geometric coefficient of variation was not calculable as more than one-third of the values were LTR.
  Week 2: number analyzed (Participants) | 45
  Week 2 | 55.5 (89.1)
  Week 4: number analyzed (Participants) | 42
  Week 4 | 63.6 (69.4)
  Week 8: number analyzed (Participants) | 43
  Week 8 | 64.4 (83.7)
  Week 16: number analyzed (Participants) | 33
  Week 16 | 78.2 (68.0)
  Week 24: number analyzed (Participants) | 32
  Week 24 | 62.7 (141.4)
  Early Termination: number analyzed (Participants) | 6
  Early Termination | 4.92 (1070.9)
  Unscheduled predose: number analyzed (Participants) | 2
  Unscheduled predose | 0.500 (NA) — Geometric coefficient of variation was not calculable as more than one-third of the values were LTR.
  Unscheduled postdose: number analyzed (Participants) | 1
  Unscheduled postdose | 0.500 (NA) — Geometric coefficient of variation was not calculable as more than one-third of the values were LTR.

3. Secondary Outcome: Serum Concentrations of Lampalizumab (Q4W)
Description: LTR results on pre-dose sample were set to 0, and LTR results on post-dose sample were set to half of LLOQ (0.5 ng/mL).
Time Frame: Baseline (Day 1, predose and postdose), Weeks 4,8,16 and 24, early termination
Population: PK population included participants randomized to lampalizumab treatment who received at least one dose of study drug and provided at least one serum sample for determination of lampalizumab. Number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Lampalizumab Q4W
Number analyzed (Participants) | 23
ng/mL
  Day 1 (Predose): number analyzed (Participants) | 22
  Day 1 (Predose) | NA (NA) — Geometric mean and geometric coefficient of variation were not calculable as more than one-third of the values were LTR.
  Day 1 (Postdose): number analyzed (Participants) | 21
  Day 1 (Postdose) | 2.08 (NA) — Geometric coefficient of variation was not calculable as more than one-third of the values were LTR.
  Week 4: number analyzed (Participants) | 22
  Week 4 | 8.52 (114.3)
  Week 8: number analyzed (Participants) | 22
  Week 8 | 10.3 (84.1)
  Week 16: number analyzed (Participants) | 21
  Week 16 | 8.66 (88.0)
  Week 24: number analyzed (Participants) | 18
  Week 24 | 9.92 (102.0)
  Early Termination: number analyzed (Participants) | 1
  Early Termination | 14.1 (NA) — Geometric coefficient of variation was not calculable as more than one-third of the values were LTR.

4. Secondary Outcome: Percentage of Participants With Ocular Adverse Events (AEs)
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether considered related to the medicinal product, any new disease or exacerbation of an existing disease, recurrence of an intermittent medical condition, or any deterioration in a laboratory value or other clinical test. Ocular AEs are the events which are localized in the ocular region.
Time Frame: Baseline up to approximately 30 weeks
Population: Safety analysis population included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Sham Q2W | Sham Q4W | Lampalizumab Q2W | Lampalizumab Q4W
Number analyzed (Participants) | 10 | 11 | 46 | 22
percentage of participants | 60.0 | 9.1 | 63.0 | 63.6

5. Secondary Outcome: Percentage of Participants With Systemic (Non-ocular) Adverse Events
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether considered related to the medicinal product, any new disease or exacerbation of an existing disease, recurrence of an intermittent medical condition, or any deterioration in a laboratory value or other clinical test. Non-ocular AEs were the systemic events.
Time Frame: Baseline up to approximately 30 weeks
Population: Safety analysis population included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Sham Q2W | Sham Q4W | Lampalizumab Q2W | Lampalizumab Q4W
Number analyzed (Participants) | 10 | 11 | 46 | 22
percentage of participants | 40.0 | 63.6 | 52.2 | 50.0

6. Secondary Outcome: Percentage of Participants With Anti-Lampalizumab Antibodies
Description: Having treatment-induced anti-drug antibodies (ADAs) was defined as being ADA-negative at baseline and ADA-positive at any post-baseline timepoint. Having treatment-enhanced ADAs was defined as being ADA-positive at baseline with titer values increased by 0.6 titer units at any post-baseline timepoint.
Time Frame: Baseline up to approximately 30 weeks
Population: Safety analysis population included all randomized participants who received at least one dose of study drug. Number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Number; unit: percentage of participants
Arm/Group | Sham Q2W | Sham Q4W | Lampalizumab Q2W | Lampalizumab Q4W
Number analyzed (Participants) | 10 | 11 | 46 | 22
percentage of participants
  Treatment-induced ADA: number analyzed (Participants) | 10 | 11 | 45 | 22
  Treatment-induced ADA | 0 | 0 | 1 | 1
  Treatment-enhanced ADA: number analyzed (Participants) | 10 | 11 | 45 | 22
  Treatment-enhanced ADA | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 30 weeks
Description: Safety analysis population included all randomized participants who received at least one dose of study drug.
Arm/Group | Lampalizumab Q2W | Lampalizumab Q4W | Sham Q2W | Sham Q4W
All-Cause Mortality (participants affected / at risk) | 2/46 | 0/22 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 7/46 | 3/22 | 0/10 | 1/11
Other Adverse Events (participants affected / at risk) | 21/46 | 13/22 | 7/10 | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lampalizumab Q2W (N=46) | Lampalizumab Q4W (N=22) | Sham Q2W (N=10) | Sham Q4W (N=11)
Scleritis (Eye disorders) | 1 | 0 | 0 | 0
Uveitis (Eye disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Non-hodgkins lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lampalizumab Q2W (N=46) | Lampalizumab Q4W (N=22) | Sham Q2W (N=10) | Sham Q4W (N=11)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 12 | 6 | 3 | 1
Eye pain (Eye disorders) | 6 | 3 | 0 | 0
Vitreous floaters (Eye disorders) | 3 | 2 | 1 | 0
Vitreous detachment (Eye disorders) | 2 | 3 | 0 | 0
Cataract subcapsular (Eye disorders) | 1 | 0 | 0 | 1
Photopsia (Eye disorders) | 1 | 0 | 1 | 0
Posterior capsule opacification (Eye disorders) | 1 | 0 | 1 | 0
Retinal haemorrhage (Eye disorders) | 1 | 0 | 1 | 0
Borderline glaucoma (Eye disorders) | 0 | 0 | 1 | 0
Cataract nuclear (Eye disorders) | 0 | 0 | 0 | 1
Conjunctival oedema (Eye disorders) | 0 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 1 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 1 | 0
Neovascular age-related macular degeneration (Eye disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 3 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 4 | 3 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0
Device breakage (Product Issues) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-24): https://cdn.clinicaltrials.gov/large-docs/59/NCT02288559/Prot_SAP_000.pdf